CLINICAL TRIAL: NCT00991458
Title: Study of Cyclosporine in Post-LASIK Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 192371-018
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Results first posted 2013-07-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Laser In Situ Keratomileusis
MeSH Terms: interventions — Cyclosporine; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cyclosporine 0.010% eye drops (Experimental): Cyclosporine 0.010% eye drops administered as 1 drop to each eye twice daily (morning and evening) for at least 2 weeks prior to LASIK surgery and up to 7 months post-LASIK surgery.
  Interventions: Drug: Cyclosporine 0.010% eye drops
- Cyclosporine 0.005% eye drops (Experimental): Cyclosporine 0.005% eye drops administered as 1 drop to each eye twice daily (morning and evening) for at least 2 weeks prior to LASIK surgery and up to 7 months post-LASIK surgery.
  Interventions: Drug: Cyclosporine 0.005% eye drops
- Placebo (Vehicle for Cyclosporine) (Placebo Comparator): Placebo eye drops administered as 1 drop to each eye twice daily (morning and evening) for at least 2 weeks prior to LASIK surgery and up to 7 months post-LASIK surgery.
  Interventions: Drug: Placebo (Vehicle for Cyclosporine)

INTERVENTIONS:
Drug: Cyclosporine 0.010% eye drops — Cyclosporine 0.010% eye drops administered as 1 drop to each eye twice daily (morning and evening) for at least 2 weeks prior to LASIK surgery and up to 7 months post-LASIK surgery.
  Arms: Cyclosporine 0.010% eye drops
Drug: Cyclosporine 0.005% eye drops — Cyclosporine 0.005% eye drops administered as 1 drop to each eye twice daily (morning and evening) for at least 2 weeks prior to LASIK surgery and up to 7 months post-LASIK surgery.
  Arms: Cyclosporine 0.005% eye drops
Drug: Placebo (Vehicle for Cyclosporine) — Placebo eye drops administered as 1 drop to each eye twice daily (morning and evening) for at least 2 weeks prior to LASIK surgery and up to 7 months post-LASIK surgery.
  Arms: Placebo (Vehicle for Cyclosporine)

SUMMARY:
This study will evaluate the safety and efficacy of Cyclosporine 0.005% and 0.010% eye drops administered twice daily before and following LASIK surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled for bilateral LASIK surgery
* Patient is in good general health
* Eye glasses prescription of -1 to -8

Exclusion Criteria:

* Significant Dry Eye
* Presence of eye disease
* Uncontrolled systemic disease
* Previous use of RESTASIS®

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 621 (Actual)
Dates: Start 2009-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Overland Park, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cyclosporine 0.010% Eye Drops | Cyclosporine 0.005% Eye Drops | Placebo (Vehicle for Cyclosporine)
Started | 207 | 209 | 205
Completed | 187 | 181 | 180
Not Completed | 20 | 28 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclosporine 0.010% Eye Drops | Cyclosporine 0.005% Eye Drops | Placebo (Vehicle for Cyclosporine) | Total
Number analyzed (Participants) | 207 | 209 | 205 | 621
Age, Customized [Number; unit: Participants]
  <30 years | 68 | 69 | 77 | 214
  30 to 40 years | 110 | 97 | 92 | 299
  >40 years | 29 | 43 | 36 | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 118 | 105 | 338
  Male | 92 | 91 | 100 | 283

OUTCOME MEASURES:

1. Primary Outcome: Time to Cure
Description: Time to cure is defined as the number of days after laser in situ keratomileusis (LASIK) surgery that the patient has corneal sensitivity (the capability of the cornea to respond to stimulation) ≥ 50 millimeters in all 9 regions of both eyes after LASIK surgery. A patient is considered cured at the first of 2 consecutive visits meeting these criteria. The Inter-Quartile Range presented is actually the 25th Quantile and the 75th Quantile obtained from the Kaplan-Meier Model.
Time Frame: 6 Months
Population: Modified Intent to Treat: all randomized and treated patients with both eyes having Post-LASIK surgery and corneal sensitivity measurements of < 25 mm in the 3 central regions at Post-Surgery Week 1.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Cyclosporine 0.010% Eye Drops | Cyclosporine 0.005% Eye Drops | Placebo (Vehicle for Cyclosporine)
Number analyzed (Participants) | 150 | 142 | 139
Days | 189.0 [181.0 to NA] — The upper limit was not reached at 6 months. | 194.0 [181.0 to 196.0] | 189.0 [180.0 to NA] — The upper limit was not reached at 6 months.

2. Secondary Outcome: Time to Worst Outcome Post-LASIK Surgery in Tear Film Assessment
Description: The time to the worst outcome post-LASIK surgery in tear film stability is assessed using the Ocular Scatter Index (OSI). The OSI is calculated by an instrument which takes images of the eye over time. OSI values ≥3.0 indicate lower tear film quality resulting in a loss of visual acuity. The worst outcome post-LASIK surgery is defined as the shortest time to OSI ≥3 across both eyes and post-LASIK surgery months 3 to 6.
Time Frame: Months 3 to 6
Population: Intent to Treat population: all randomized patients for whom data are available for this outcome measure.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cyclosporine 0.010% Eye Drops | Cyclosporine 0.005% Eye Drops | Placebo (Vehicle for Cyclosporine)
Number analyzed (Participants) | 177 | 173 | 174
Seconds | 11.2 (4.24) | 12.0 (4.51) | 11.5 (4.39)

3. Secondary Outcome: Percentage of Patients With Cumulative Poor Vision
Description: Cumulative Poor Vision is determined binocularly per patient (using both eyes at the same time) from the Poor Vision question on the Ocular Surface Disease Index (OSDI) questionnaire. Severity of poor vision is graded on a 5-point scale (0 = none of the time, 1 = some of the time, 2 = half of the time, 3 = most of the time, 4 = all of the time). Cumulative poor vision is defined as at least one poor vision score ≥ 1 beginning at Month 3 post-LASIK.
Time Frame: Month 3, Month 4, Month 5, Month 6
Population: Intent to treat: all randomized patients.
Measure: Number; unit: Percentage of Patients
Arm/Group | Cyclosporine 0.010% Eye Drops | Cyclosporine 0.005% Eye Drops | Placebo (Vehicle for Cyclosporine)
Number analyzed (Participants) | 207 | 209 | 205
Percentage of Patients
  Month 3 | 15.0 | 18.7 | 19.0
  Month 4 | 17.9 | 22.5 | 23.9
  Month 5 | 21.7 | 26.3 | 24.9
  Month 6 | 23.7 | 26.8 | 26.3

4. Secondary Outcome: Worst Outcome Post-LASIK Surgery in Reading Speed Assessment
Description: Reading speed is determined using the MNREAD™ Reading Card. The MNREAD™ reading card is designed to simulate a normal every day reading scenario using binocular vision (both eyes at the same time). The MNREAD™ Reading speed is calculated as (60) X [Number of words on card - (reading errors)]/ (number of seconds until the card is read). The worst outcome is defined as the smallest number of words per minute across post-LASIK surgery months 3 to 6.
Time Frame: Months 3 to 6
Population: Intent to Treat population: all randomized patients for whom data are available for this outcome measure.
Measure: Mean (Standard Deviation); unit: Words Per Minute (WPM)
Arm/Group | Cyclosporine 0.010% Eye Drops | Cyclosporine 0.005% Eye Drops | Placebo (Vehicle for Cyclosporine)
Number analyzed (Participants) | 206 | 209 | 205
Words Per Minute (WPM) | 173.0 (40.17) | 173.7 (42.18) | 167.4 (45.21)

ADVERSE EVENTS:
Arm/Group | Cyclosporine 0.010% Eye Drops | Cyclosporine 0.005% Eye Drops | Placebo (Vehicle for Cyclosporine)
Serious Adverse Events (participants affected / at risk) | 2/207 | 0/209 | 3/205
Other Adverse Events (participants affected / at risk) | 78/207 | 66/209 | 66/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cyclosporine 0.010% Eye Drops (N=207) | Cyclosporine 0.005% Eye Drops (N=209) | Placebo (Vehicle for Cyclosporine) (N=205)
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Haemorrhagic Ovarian Cyst (Reproductive system and breast disorders) | 1/115 | 0/118 | 0/105
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/115 | 0/118 | 1/105
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/115 | 0/118 | 1/105
Refraction Disorder (Eye disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine 0.010% Eye Drops (N=207) | Cyclosporine 0.005% Eye Drops (N=209) | Placebo (Vehicle for Cyclosporine) (N=205)
Dry Eye (Eye disorders) | 52 | 48 | 47
Punctate Keratitis (Eye disorders) | 13 | 11 | 10
Vision Blurred (Eye disorders) | 13 | 7 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.